CLINICAL TRIAL: NCT06120036
Title: Dosing and Tolerability of Deoxycholic Acid Versus Polidocanol in the Treatment of Neurofibromatosis Type 1 Cutaneous Neurofibromas
Brief Title: Dosing and Tolerability of Deoxycholic Acid vs. Polidocanol in the Treatment of Neurofibromatosis Type 1 Cutaneous Neurofibromas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Director, Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022P001946
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Neurofibromatosis 1
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Deoxycholic Acid; Polidocanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Kybella Injection (Active Comparator)
  Interventions: Drug: Kybella
- Asclera Injection (Active Comparator)
  Interventions: Drug: Asclera

INTERVENTIONS:
Drug: Kybella — Injection into the cutaneous Neurofibromas lesion.
  Arms: Kybella Injection
Drug: Asclera — Injection into the cutaneous Neurofibromas lesion.
  Arms: Asclera Injection

SUMMARY:
This study will evaluate the tolerability and effectiveness of two treatments in Neurofibromatosis Type 1 Cutaneous Neurofibromas. These treatments are: Kybella and Asclera injection. Each patient will have a treatment and a control site.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females ≥18 years of age
2. Have a diagnosis of NF1 based on germline genetic testing or by meeting ≥ 2 the following criteria:

   1. Family history of NF1
   2. Six or more light brown ("cafe-au-lait") spots on the skin
   3. Presence of two or more neurofibromas of any type, or one or more plexiform neurofibromas
   4. Freckling under the arms or in the groin area
   5. Two or more pigmented, benign bumps on the eye's iris (Lisch nodules)
   6. A distinctive bony lesion: dysplasia (abnormal growth) of the sphenoid bone behind the eye, or dysplasia of long bones, often in the lower leg
   7. Tumor on the optic nerve that may interfere with vision
3. Patients must be seeking treatment for cNF
4. Patients must have ≥ 6 paired cNF per modality (3 treated and 3 untreated). cNF should be visible and measure between 2-8mm in size. These must be in areas amenable to treatment and surveillance with digital photography.
5. cNF must be located on the trunk, arms or legs of the patient
6. Able and willing to comply with all visit, treatment and evaluation schedules and requirements
7. Able to understand and provide written informed consent

Exclusion Criteria:

1. Patients who are undergoing other treatment modalities or investigational agents for their cNF lesions
2. Individuals who cannot give informed consent or adhere to study schedule
3. Actively tanning during the course of the study
4. Adverse reactions to compounds of any external agent (e.g., gels, lotions or anesthetic creams) required for use in the study, if no alternative to the said agent exists;
5. Known allergy to injectable anesthetics, polidocanol or deoxycholic acid
6. Those with acute thromboembolic diseases
7. Those with bleeding abnormalities or those who are currently being treated with antiplatelet or anticoagulant therapy
8. Those with dysphagia
9. Women who are pregnant
10. Any condition which, in the Investigator's opinion, would make it unsafe (for the participant or study personnel) to treat the participant as part of this research study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 3 months after treatment
  Device based treatment will be considered tolerable if <40% of participants treated have a >grade 2 adverse event (AE). A grade 2 AE is defined as an adverse event that requires treatment.

SECONDARY OUTCOMES:
Treatment specific patient reported outcomes (PRO) | Baseline, 1 day after treatment, 1 week after treatment, 1 month after treatment, 2 months after treatment, 3 months after treatment, 6 months after treatment, 12 months after treatment
  NRS11, modality specific satisfaction assessment
Clinician reported outcomes (ClinRO) | Baseline, 3 months after treatment, 6 months after treatment, 12 months after treatment
  Clinician assessment of cNF via questionnaire. Physician rates degree of change of treated and control cNFs on a scale from -3 (no change) to 3 (very large improvement).
Modified SkinDex for cNF | Baseline, 3 months after treatment, 6 months after treatment, 12 months after treatment
  Health-related quality of life measure. Asks how much participants have been bothered by cNFs over the past week from 0 (never bothered) to 5 (always bothered).

OTHER OUTCOMES:
Rate of healing | Baseline, 3 months after treatment, 6 months after treatment, and 12 months after treatment
  Measured clinically via photography completed by a member of the study team at baseline, 3-month, 6-month, and 12-month post-treatment.
cNF appearance | Baseline, 3 months after treatment, 6 months after treatment, and 12 months after treatment
  Clinically completed 2D and 3D photography Cherry Imaging.
Biologic effect | 3 months after treatment
  Degree of tissue necrosis on skin lesion biopsy at 3 months as assessed by review of area of necrosis in histology slides.

CONTACTS AND LOCATIONS:
Overall Officials: Richard R Anderson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Wellman Center for Photomedicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No